CLINICAL TRIAL: NCT06562907
Title: A Phase 1 Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Single Ascending Oral Doses of GS-4571 in Healthy Participants, Multiple Ascending Oral Doses of GS-4571 in Nondiabetic Obese Participants and Nonobese Participants With Type 2 Diabetes Mellitus (T2DM), and to Evaluate the Effect of Food and an Acid-Reducing Agent on Pharmacokinetics of GS-4571
Brief Title: Study of GS-4571 in Healthy Participants, Nondiabetic Obese Participants, and Nonobese Participants With Type 2 Diabetes Mellitus (T2DM)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-506-6610
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Weight Management
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A Single-ascending Dose (SAD) in Healthy Participants (Experimental): Participants will be randomized into 4 + (optional) 1 dose escalating cohorts and will receive GS-4571 or placebo to match (PTM) GS-4571 on Day 1, to determine the maximum tolerated dose:
  * Cohort 1: Dose 1 GS-4571, administered orally as a single dose, in a fasting state.
  * Cohort 2: Dose 2 GS-4571, administered orally as a single dose, in a fasting state.
  * Cohort 3: Dose 3 GS-4571, administered orally as a single dose, in a fasting state.
  * Cohort 4: Dose 4 GS-4571, administered orally as a single dose, in a fasting state.
  * Cohort 5 (optional): Dose 5 GS-4571, administered orally as a single dose, in a fasting state.
  Interventions: Drug: GS-4571; Drug: Placebo
- Part B Food/PPI Effect in Healthy Participants (Experimental): Participants will be randomized into 2 sequence groups in Cohort 6 and will receive the highest dose found to be safe and well tolerated in Part A of GS-4571 and omeprazole. The two sequential groups will receive the following treatments:
  * Treatment A: Up to the highest single dose of GS-4571 evaluated in Part A, fasting.
  * Treatment B: Up to the highest single dose of GS-4571 evaluated in Part A, nonfasting (high-fat/high-calorie meal).
  * Treatment C (optional): Omeprazole, once-daily (QD) for 5 days, fasting.
  * Treatment D (optional): Omeprazole followed by up to the highest single dose of GS-4571 evaluated in Part A, 2 hours later, fasting.
  Interventions: Drug: GS-4571; Drug: Omeprazole
- Part C Multiple-ascending Dose (MAD) in Nondiabetic Obese Participants (Experimental): Participants randomized in Cohorts 7-9 will be randomized to receive up to 4 escalating doses of GS-4571 or PTM QD for 12 weeks, as follows:
  * Cohort 7: Up to dose determined from Part A of GS-4571 or PTM in obese participants, QD, in a non-fasting state
  * Cohort 8: Up to 3-fold the Cohort 7 dose of GS-4571 or PTM in obese participants, QD, in a non-fasting state
  * Cohort 9: Up to 2-fold the Cohort 8 dose of GS-4571 or PTM in obese participants, QD, in a non-fasting state
  * Cohort 10 is optional and will receive GS-4571 or PTM QD for 12 weeks in case it is opened for enrollment as follows:
    * Up to 2-fold the Cohort 9 dose of GS-4571 or PTM in obese participants, QD, in a non-fasting state.
  Interventions: Drug: GS-4571; Drug: Placebo
- Part D Multiple Dose in Nonobese Participants With T2DM (Experimental): Participants randomized in Cohort 11 will receive up to the highest dose of GS-4571 or PTM in T2DM, QD, in a non-fasting state for 12 weeks.
  Interventions: Drug: GS-4571; Drug: Placebo

INTERVENTIONS:
Drug: GS-4571 — Administered orally
Drug: Placebo — Administered orally
  Arms: Part A Single-ascending Dose (SAD) in Healthy Participants; Part C Multiple-ascending Dose (MAD) in Nondiabetic Obese Participants; Part D Multiple Dose in Nonobese Participants With T2DM
Drug: Omeprazole — Administered orally
  Arms: Part B Food/PPI Effect in Healthy Participants

SUMMARY:
The goal of this clinical study is to learn more about the study drug, GS-4571, and how safe it is in 3 groups, i) Healthy participants, ii) Healthy non-diabetic obese participants, and iii) Non-obese participants with Type 2 Diabetes Mellitus (T2DM).

The primary objectives of this study are:

* To characterize the pharmacokinetics (PK) of GS-4571 following single and multiple ascending oral doses of GS-4571.
* To evaluate the effect of concomitant food intake and (if conducted) a representative acid-reducing agent (proton pump inhibitor (PPI), omeprazole) on the PK of GS-4571.
* To evaluate the safety and tolerability of single and multiple ascending oral doses of GS-4571.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals must be glucagon-like peptide-1 receptor agonist (GLP-1RA) naïve OR last dose was at least 6 months prior to screening.
* Part A (SAD) and Part B (Food/PPI Effect): eligible individuals in Cohorts 1-4, (optional cohort 5) and 6 will include healthy individuals with BMI of ≥ 19 and < 30 kg/m^2, and no significant medical history.

Individuals will also be in good general health as determined by the investigator at the screening evaluation performed no more than 28 days prior to the scheduled first dose.

* Part C (MAD in nondiabetic obese individuals): Eligible individuals in Cohorts 7-9 and (optional cohort 10) will be individuals with obesity with BMI ≥ 30 kg/m^2 and < 45 kg/m^2 with a total body weight > 50 kg, and nondiabetic (HbA1c < 6.5%). Eligible individuals will also be individuals with stable body weight (< 5% change) for 90 days prior to screening visit based on individual report.
* Part D (multiple doses in non-obese T2DM): eligible individuals in Cohort 11 will be individuals with T2DM HbA1c ≥ 7.0% and ≤ 10.5% with BMI of ≥ 19 and < 30 kg/m^2 and treated with diet and/or exercise, and/or metformin monotherapy.

Key Exclusion Criteria:

* Have any serious or active medical or psychiatric illness (including depression) that, in the opinion of the investigator, would interfere with individual treatment, assessment, or compliance with the protocol. This would include acute pancreatitis, or history of pancreatitis, acute gallbladder disease, and renal, cardiac, hematological, hepatic, pulmonary (including chronic asthma), endocrine (including diabetes [with the exception of T2DM for individuals included in Part D only]), central nervous, gastrointestinal (including an ulcer), vascular, metabolic (thyroid disorders, adrenal disease), immunodeficiency disorders, active infection, or malignancy that are clinically significant or requiring treatment.
* Current symptoms of diabetic retinopathy or examination indicating diabetic retinopathy within one year of screening.
* Any electrolyte disturbances identified at screening considered to be clinically significant in the opinion of the investigator (eg, hypokalemia, hypocalcemia, or hypomagnesemia).
* Any condition that could lead to electrolyte disturbances (eg, eating disorder) in the opinion of the investigator.
* History of syncope, palpitations, or unexplained dizziness.
* Active, or history of, significant cardiac disease or conduction abnormality
* History of implanted defibrillator or pacemaker.
* Have been treated with the following within 6 months prior to screening or is expected to receive these agents during the study: GLP-1RAs, systemic steroids, immunosuppressant therapies, or chemotherapeutic agents (eg, corticosteroids, immunoglobulins, other immune or cytokine-based therapies).
* Previously stopped use of GLP-1RAs secondary to severe side effects including nausea, constipation, diarrhea, or emesis.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Single-Dose PK Parameter AUCinf of GS-4571 | Up to 96 hours postdose
  AUCinf is defined as area under the concentration versus time curve extrapolated to infinite time.
Single-Dose PK Parameter Cmax of GS-4571 | Up to 96 hours postdose
  Cmax is defined as the maximum observed concentration of drug in plasma.
Multiple-Dose Plasma PK Parameter: AUCtau of GS-4571 | Up to 96 hours postdose
  AUCtau is defined as area under the concentration versus time curve over the dosing interval.
Multiple-Dose Plasma PK Parameter: Cmax of GS-4571 | Up to 96 hours postdose
  Cmax is defined as the maximum observed concentration of drug in plasma.
Percentage of Participants of Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), or Deaths | Day 1 up to 95 days
Percentage of Participants of Treatment-Emergent Laboratory Abnormalities | Day 1 up to 95 days

SECONDARY OUTCOMES:
Percentage Change From Baseline (CFB) in Body Weight in Nondiabetic Obese Participants | Day 1 up to 95 days

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (2):
- United States (2):
  - ICON Early Phase Services, LLC, San Antonio, Texas
  - ICON, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06562907